CLINICAL TRIAL: NCT04659902
Title: The Influence of Protein Form and the Presence or Absence of Calcium on Gut Hormone Secretion and Gastric Emptying in Lean Healthy Individuals
Brief Title: Protein, Calcium and Gut Hormone Secretion
Acronym: PROCAL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Principal Investigator, Jonathan Watkins, PhD Research Programme in Health, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PROCAL2-JW
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: There are 4 conditions where participants will ingest different forms of protein in the presence or absence of calcium.
Who Masked: Participant, Investigator
Masking Description: Participant will not be told which drink they will ingest until the end of the study.
  Individuals not collaborating on the study will randomise the drink order and make up the drinks so the investigator is blinded to which drink the participant will ingest.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CON (Placebo Comparator): Participants will ingest a drink containing a control protein only
  Interventions: Dietary Supplement: Protein form
- CON-C (Active Comparator): Participants will ingest a drink containing a control protein plus Capolac® (9547 mg to provide 2500mg of calcium)
  Interventions: Dietary Supplement: Protein form
- PRO (Active Comparator): Participants will ingest a drink containing an aggregate protein only
  Interventions: Dietary Supplement: Protein form
- PRO-C (Active Comparator): Participants will ingest a drink containing an aggregate protein plus Capolac® (9547 mg to provide 2500mg of calcium)
  Interventions: Dietary Supplement: Protein form

INTERVENTIONS:
Dietary Supplement: Protein form — Protein form and absence or presence of calcium manipulated

SUMMARY:
Hormones that are produced by our stomach and intestines play a role in regulating our appetite and health, and are therefore of high interest for managing conditions such as obesity and Type 2 Diabetes (T2D). Two important hormones, called GLP-1 and PYY, are released from the same intestinal cell. The food we eat influences the release of these hormone and evidence suggests that protein and calcium are key nutrients that stimulate the secretion of GLP-1, while the influence of this combination on PYY release is less clear. Furthermore, gastric emptying affects the rate of absorption of nutrients and by manipulating the structural form of protein, in the absence or presence of calcium, we may be able to learn more about the processes mediating the gut hormone response. We hypothesise that gut hormone secretion will be enhanced following the ingestion of a partially digested protein in the presence of calcium versus a control protein without calcium. Additionally, the ingestion of the partially digested protein will result in faster gastric emptying compared to the control protein.

DETAILED DESCRIPTION:
Recent work at the University of Bath has shown that when ingested with 50 g whey protein hydrolysate, Capolac® (milk minerals high in calcium) potently stimulates availability of the important hormone glucagon-like peptide-1 (GLP-1). However, it is currently unclear how the form of protein ingested with the presence or absence of calcium may affect gut hormone secretion and gastric emptying. Therefore we aim to perform a study on the effect of co-ingesting two different forms of protein in the presence or absence of calcium on gut hormone availability and gastric emptying. This project will help provide key evidence to aid future work and recommendations for nutrition-based interventions for the prevention and management of obesity and T2D.

Fifteen metabolically healthy men and women, age 18-65 years, BMI between 18.5 and 25 kg/m2 will be recruited to participate in a randomised crossover study. Each participant will undergo 4 trials. Each trial will last ~3 hours and will be separated by a minimum of 48h:

CONTROL (CON) - 30 g Control protein only CONTROL + CALCIUM (CON-C) - 30 g Control protein + 9547 mg Capolac® (2500 mg of calcium ingested) PROTEIN (PRO) - 30 g Aggregate protein only PROTEIN + CALCIUM (PRO-C) - 30 g Aggregate protein + 9547 mg Capolac® (2500 mg of calcium ingested)

Each of these drinks will also contain 500 mL of water, low calorie sweetener (80 mg sucralose) and will be labelled with 150 mg 13C1 sodium acetate, and 100 mg 13C1 sodium octanoate for the measurement of gastric emptying.

Participants will be asked to arrive to the laboratory between 09:00 and 10:00 am after not eating for between 10-14 hours i.e. in a fasted state (water intake is permitted and encouraged). Upon arrival at the laboratory a trained phlebotomist staff member will insert a cannula (a small plastic tube) into a pre-heated dorsal hand vein on the back of the hand, or if unsuccessful, the antecubital vein. Participants will then be given one of the four test drinks, which once ingested will initiate the trial. Just after the ingestion of the test drink we will ask participants to fill out a palatability scale.

Blood samples will be taken at baseline, and at 15, 30, 45, 60, 90, and 120 minutes after ingestion of the test drink. Breath samples will be collected in exetainers at baseline, and every 5 minutes until the 120-minute time point to determine gastric emptying. An appetite questionnaire will also be completed at baseline and every 60 minutes after ingestion of the test drink to assess appetite sensations. After the 120-minute time point participants will be asked to consume a lunch meal until they are comfortably full. Once satisfied with the lunch meal they will fill out the final appetite questionnaire. The trial day will then be complete. Following study completion participants will be asked to complete a restrained eating questionnaire.

A subset of 5 participants will be fitted with a nasogastric tube by a qualified BAPEN nurse. 5ml aspirate from the stomach will be samples at baseline, 30, 60, and 120 minutes which will be distributed equally for analyte profiling and in vitro culture work. 3 ml gastric aspirate will be used to stimulate a GLUTag cell line. Experiments will be performed by incubating cells with the neutralised gastric aspirate in 250 µl Krebs Ringer Buffer (KRB) for 2 h at 37˚C, 5 % CO2. A second culture, identical to that previously described will be conducted, only with the addition of specific cell receptor antagonists.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5-25.0 kg∙m-2
* Age 18-65 years
* Able and willing to provide informed consent and safely comply with study procedures
* Females to maintain record of regular menstrual cycle phase or contraceptive use
* No anticipated changes in diet/physical activity during the study (e.g. holidays or diet plans)

Exclusion Criteria:

* Allergies or adverse reactions to calcium or milk proteins.
* Contradictions to a high intake of calcium e.g. history of kidney stones
* Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias
* Any diagnosed gastrointestinal or metabolic disease (e.g. type 1 or type 2 diabetes)
* Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment
* Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)
* Any reported recent (<6 months) change in body mass (± 3%)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
incremental area under the curve (iAUC) for total plasma GLP-1 | 2 hours
  Blood sampling

SECONDARY OUTCOMES:
Gastric emptying | 2 hours
  gastric emptying measured via acetate breath test
in vitro gut hormone secretion | 2 hours
  GLP-1 and peptide tyrosine tyrosine (PYY) secretion from GLUTag cell line
iAUC for total PYY | 2 hours
  Blood sampling
iAUC for plasma and gastric amino acid profile | 2 hours
  blood and gastric sampling
iAUC for plasma Dipeptidyl Peptidase-IV (DPP4) | 2 hours
  blood sampling
iAUC for plasma insulin | 2 hours
  blood sampling
iAUC for plasma glucose | 2 hours
  blood sampling
iAUC for active plasma GLP-1 | 2 hours
  blood sampling
Visual appetite scales | 2 hours
  4 questions to measure subjective appetite, hunger, fullness and prospective consumption, participant marks where they feel they are on a continuum from one extreme to another e.g. i have never been so hungry to i have never been more hungry
ad libitum lunch meal | 2 hours
  a pasta lunch meal is provided where the participant eats as much as they want until they are comfortably full, energy intake is measured

CONTACTS AND LOCATIONS:
Locations (1):
- Department For Health, University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watkins JD, Smith HA, Hengist A, Nielsen SB, Mikkelsen UR, Saunders J, Koumanov F, Betts JA, Gonzalez JT. Effects of physical form of beta-lactoglobulin and calcium ingestion on GLP-1 secretion, gastric emptying and energy intake in humans: a randomised crossover trial. Br J Nutr. 2024 May 28;131(10):1730-1739. doi: 10.1017/S0007114524000321. Epub 2024 Jan 30. PMID 38287700